CLINICAL TRIAL: NCT01912300
Title: Nutritional Adaptation to Contemporary Sedentary Behaviors and Physical Exercise in Youth: Effect of Weight Status
Brief Title: Nutritional Adaptations to Physical or Sedentary Activities in Youth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Université Blaise Pascal, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, THIVEL David, PhD scientist, Université Blaise Pascal, Clermont-Ferrand
Other Study IDs: AU1033
Record Dates: First submitted 2013-07-10; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Passive Video Games (PVG); Active Video Games (AVG); Exercise (EX)
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean adolescents (Experimental)
  Interventions: Behavioral: experimental condition: Passvice Video game; Avtive Video game; Exercise
- Obese adolescents (Experimental)
  Interventions: Behavioral: experimental condition: Passvice Video game; Avtive Video game; Exercise

INTERVENTIONS:
Behavioral: experimental condition: Passvice Video game; Avtive Video game; Exercise

SUMMARY:
Sedentary behaviors have been shown to increase food consumption among youth and adults. The recent active video games devices have been suggested to compensate for the increased energy intake they induce by the increased energy expenditure they generate. To date no study has been conducted to question whether or not such modern sedentary activities induce energy consumption modification in youth. The aim of this work is to compare the impact of a passive video games vs. active video games vs. physical exercise in terms of subsequent energy intake and appetite feelings in normal weight and obese youth.

DETAILED DESCRIPTION:
After a medical inclusion, the adolescents will have to realise a DXA to assess their body composition and a submaximal exercise to evaluate their aerobic capacities.

They will have then to enter the laboratory on three different occasions in a randomized order from 8am to 730pm: At 8am they will receive a calibrated breakfast. then, at 1045; they will have to complete one of the experimental condition: 1) one hour of passive video game; 2) one hour of active video game; 3) a cycling exercise. at 1215 and 0630pm, they will be offered ad libitum meals. At regular intervals through the day, their appetite feelings will be assessed using Visual analogue scales.

Energy expenditure will be assessed thanks to cardiofrequencemeters during the 1h PVG and and by indirect calomitery (K4b2) during the active video game.

Ad libitum energy consumption will be assessed by investigators and recorded for each participants.

ELIGIBILITY:
Inclusion Criteria:

* male
* 12-15 years old
* BMI defining obesity (Cole et al., 2000)
* Not being under diet restriction
* Information and consent forms have to be signed by the adolescent and his legal representative
* being registered to the national social security system

Exclusion Criteria:

* Being under medication
* contraindication to exercise
* smokers
* dieting

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
ad libitum energy intake in kcal during the different experimental sessions: AVG, PVG and EX | up to 2 months
  At lunch and iner time on AVG, PVG and EX (the 3 experimental sessions), an ad libitum buffet meal will be oofered to the participants and their energy consumption will be weighted and registered by the investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory AME2P, Aubière, France